CLINICAL TRIAL: NCT02519023
Title: Transversus Abdominis Plane (TAP) Infiltration vs. Surgical Infiltration of Local Anesthetic in Laparoscopic and Robotic Assisted Hysterectomy
Brief Title: TAP vs Surgical Infiltration of Local Anesthetic in Laparoscopic and Robotic Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7152222222
Record Dates: First submitted 2015-07-28; First posted 2015-08-10 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-01

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine; Ultrasonography; Epinephrine; Acetaminophen; Ibuprofen; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP-Block with liposomal bupivacaine (Experimental): TAP infiltration will contain 10 mL of 0.25 % bupivacaine with epinephrine injected followed by 20 mL of a 50:50 mixture of liposomal bupivacaine and normal saline. This will then be repeated on the contralateral side. In the same arm the surgeon infiltration into the incision will consist of 10 ml of normal saline per port site, 5 ml prior to incision and 5 ml prior to closure at each port site.
  Interventions: Drug: Liposomal Bupivacaine; Device: Ultrasound; Drug: Epinephrine; Drug: acetaminophen; Drug: ibuprofen; Drug: Oxycodone
- Surgical infiltration with bupivacaine (Active Comparator): Surgical Infiltration of the study solution will be performed both prior to incision and at the end of surgery just prior to closure of incisions. At each time, the surgeon will inject 5 mL of 0.25% bupivacaine into each of the port site incisions.
  Interventions: Drug: Bupivacaine; Device: Ultrasound; Drug: acetaminophen; Drug: ibuprofen; Drug: Oxycodone

INTERVENTIONS:
Drug: Liposomal Bupivacaine — In one arm the TAP infiltration will contain 10 mL of 0.25 % bupivacaine with epinephrine injected followed by 20 mL of a 50:50 mixture of liposomal bupivacaine and normal saline. This will then be repeated on the contralateral side.
  Other Names: Exparel
  Arms: TAP-Block with liposomal bupivacaine
Drug: Bupivacaine — Surgical Infiltration of the study solution will be performed both prior to incision and at the end of surgery just prior to closure of incisions. At each time, the surgeon will inject 5 mL of 0.25% bupivacaine into each of the port site incisions.
  Arms: Surgical infiltration with bupivacaine
Device: Ultrasound — An ultrasound, which is a beam of high frequency sound that allows one to visualize images in the body, will be used to aid investigators to observe the local anesthetic being infiltrated into the plane
Drug: Epinephrine — TAP infiltration will contain 10 mL of 0.25 % bupivacaine with epinephrine.
  Arms: TAP-Block with liposomal bupivacaine
Drug: acetaminophen — all individuals will receive scheduled acetaminophen (1 gram every 6 hours),
Drug: ibuprofen — all individuals will receive scheduled ibuprofen (800 mg every 8 hours)
Drug: Oxycodone — all individuals will receive PRN oxycodone 5-10mg q4h if pain is rated at more than 5 out of 10 on a numerical pain scale.

SUMMARY:
Laparoscopic and Robotic assisted hysterectomy is a surgical procedure that is a minimally invasive way in which to remove the uterus, which has less scarring and fewer complications. However, this procedure, much like its open-surgical counterpart, is often associated with significant post-operative pain. To augment this pain there are many different analgesic techniques available to offset pain. Ultrasound-guided transversus abdominis plane (TAP) block is one such procedure involving the injection of a local anesthetic into the plane of the transversus abdominal muscle where the terminal branches of nerves lie. A similar, yet different analgesic approach is that of direct injection of local anesthetic into the incision by the surgeon during or just after surgical procedures. These two approaches have both been proven to decrease post-operative pain in patients for many procedures, but never compared to one another.

DETAILED DESCRIPTION:
This is a double blinded randomized study. All patients will receive one form of local anesthetic pain relief either from TAP or infiltration. Patients will be randomized to one of two study arms in a double-blinded, placebo controlled study. All patients will receive a TAP infiltration and all patients will receive infiltration into the incision.

In one arm the TAP infiltration will contain 10 mL of 0.25 % bupivacaine with epinephrine injected followed by 20 mL of a 50:50 mixture of liposomal bupivacaine and normal saline. This will then be repeated on the contralateral side. In the same arm the surgeon infiltration into the incision will consist of 10 ml of normal saline per port site, 5 ml prior to incision and 5 ml prior to closure at each port site.

In the second arm the bilateral TAP infiltration will consist of 30 mL of normal saline per side. In the same arm the surgeon infiltration will consist of 10 mL of 0.25% bupivacaine per port site. The surgeon infiltration will consist of 5 ml of 0.25% bupivacaine prior to incision and 5 ml of 0.25% bupivacaine prior to closure at each port site.

A TAP infiltration is an injection of local anesthetic under the covering of the transversus abdominis muscle layer which provides effective post operative analgesia.2-5 This layer is found using an ultrasound, which is a beam of high frequency sound that allows one to visualize images in the body. Then using this ultrasound the investigators can see our needle as it pierces the covering of the transversus abdominis muscle layer and watch as the local anesthetic is infiltrated into this plane. This is done on both sides of the abdomen to provide analgesia to the skin, muscle, and facial layers of the abdomen. This is currently standard of care at our institution and will be performed within one hour of surgical incision. The injection will consist of 10 mL of 0.25% bupivacaine with epinephrine followed by 20 mL of liposomal bupivacaine saline mixture or 10 ml of saline followed by 20 ml of saline and then repeated on the contralateral side.

Surgical Infiltration of the study solution will be performed both prior to incision and at the end of surgery just prior to closure of incisions. At each time, the surgeon will inject 5 mL of 0.25% bupivacaine into each of the port site incisions.

Investigational Drug Service (IDS) pharmacy will be charged with the blinding of medications vs. saline for these procedures.

Following the procedure, all individuals will receive scheduled acetaminophen (1 gram every 6 hours), scheduled ibuprofen (800 mg every 8 hours), and PRN oxycodone 5-10mg q4h if pain is rated at more than 5 out of 10 on a numerical pain scale.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* Females >/=18-years of age
* Scheduled for laparoscopic/robot-assisted hysterectomy.

Exclusion Criteria

* Contraindication to surgical infiltration or regional blockade
* History of long term opioid intake (greater than 3 weeks prior to surgery) or chronic pain disorder
* Inability to understand the informed consent and demands of the study
* Surgery scheduled to start after 1700

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2016-07; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Geller, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feierman DE, Kronenfeld M, Gupta PM, Younger N, Logvinskiy E. Liposomal bupivacaine infiltration into the transversus abdominis plane for postsurgical analgesia in open abdominal umbilical hernia repair: results from a cohort of 13 patients. J Pain Res. 2014 Aug 16;7:477-82. doi: 10.2147/JPR.S65151. eCollection 2014. PMID 25170277
- [Background] Mitchell AU, Torup H, Hansen EG, Petersen PL, Mathiesen O, Dahl JB, Rosenberg J, Moller AM. Effective dermatomal blockade after subcostal transversus abdominis plane block. Dan Med J. 2012 Mar;59(3):A4404. PMID 22381092
- [Background] Niraj G, Searle A, Mathews M, Misra V, Baban M, Kiani S, Wong M. Analgesic efficacy of ultrasound-guided transversus abdominis plane block in patients undergoing open appendicectomy. Br J Anaesth. 2009 Oct;103(4):601-5. doi: 10.1093/bja/aep175. Epub 2009 Jun 26. PMID 19561014
- [Background] Petersen PL, Mathiesen O, Torup H, Dahl JB. The transversus abdominis plane block: a valuable option for postoperative analgesia? A topical review. Acta Anaesthesiol Scand. 2010 May;54(5):529-35. doi: 10.1111/j.1399-6576.2010.02215.x. Epub 2010 Feb 17. PMID 20175754
- [Background] Singh M, Chin KJ, Chan V. Ultrasound-guided transversus abdominis plane (TAP) block: a useful adjunct in the management of postoperative respiratory failure. J Clin Anesth. 2011 Jun;23(4):303-6. doi: 10.1016/j.jclinane.2010.05.012. PMID 21663815

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
Started | 49 | 38
Completed | 31 | 31
Not Completed | 18 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Median (Full Range); unit: years] | 58 [32 to 77] | 62 [32 to 88] | 59 [32 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Use for Pain Control
Description: total opioid used from time 0 after surgery through 72 hours after surgery was complete.
Time Frame: 72 hours
Measure: Median (Full Range); unit: mg Morphine equivalents
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
Number analyzed (Participants) | 31 | 31
mg Morphine equivalents | 20.8 [0 to 66] | 25.0 [5 to 72]

2. Secondary Outcome: Maximum Pain Scores as Measured by Numerical Pain Rating Scale (0-10)
Description: the Numerical rating scale goes from 0 (lowest) to 10 (highest). Higher values are a worse outcome. The maximal number for maximal pain scores from 0-72 hours is 30. Thus the range for this outcome is 0 to 30 with 30 being a worse outcome. This is because the 0-72 hour maximal pain scores are additive from the 0-24, 24-48, and 48-72 hours. Each 24 hour subset has a maximal score of 10 and adding all three results in maximal score of 30.
Time Frame: 0-72 hours post-procedure
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
Number analyzed (Participants) | 31 | 31
scores on a scale | 8 [0 to 29] | 13 [3 to 30]

3. Secondary Outcome: Total Opioid Taken by Patient as Tabulated and Converted to Morphine Equivalents
Time Frame: 0-24 post-procedure
Measure: Median (Full Range); unit: mg of morphine equivalents
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
Number analyzed (Participants) | 31 | 31
mg of morphine equivalents | 7.5 [0 to 55] | 22.5 [0 to 90]

4. Secondary Outcome: Quality of Recovery 15 (QoR15) Score
Description: The quality of recovery is a survey given to patients. It is 15 questions. The scale of the QOR 15 Score is 0 to 150. 150 is a better outcome.
Time Frame: 72 hours post-procedure
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
Number analyzed (Participants) | 31 | 31
scores on a scale | 126 [79 to 146] | 115 [65 to 136]

5. Secondary Outcome: Overall Benefit of Analgesia Score (OBAS)
Description: The overall benefit of analgesia score is based off 7 questions given to patients it is scored 0-28. 28 is considered a worse outcome.
Time Frame: 72 hours post-procedure
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
Number analyzed (Participants) | 31 | 31
scores on a scale | 2 [0 to 10] | 3 [0 to 11]

6. Secondary Outcome: Number of Participants With Nausea and Vomiting
Time Frame: 72 hours post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
Number analyzed (Participants) | 31 | 31
Participants | 10 | 16

7. Secondary Outcome: Length of Time in Phase 1 and Phase 2 of Recovery
Description: time from start of recovery until patient was deemed ready to discharge from phase 2 recovery. Phase 2 recovery is the phase of the post anesthesia care where patients are readied to be discharge form the post anesthesia care unit. There are guidelines with regards to when patients are able to be discharged and when those points are met by the patient they are deemed ready to discharge.
Time Frame: an expected average of 120 mins
Measure: Median (Full Range); unit: hours
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
Number analyzed (Participants) | 31 | 31
hours | 3.3 [1 to 8] | 3.1 [1 to 9]

8. Secondary Outcome: Number of Patients Admitted Post Operatively
Time Frame: 72 hours post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
Number analyzed (Participants) | 31 | 31
Participants | 11 | 16

9. Secondary Outcome: Opioid Used From 24-48 Hours Post Surgery
Description: opioids in mg of morphine equivalents used from 24-48 hours after surgery
Time Frame: 24-48 hours after the end of surgery
Measure: Median (Full Range); unit: mg of morphine equivalents
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
Number analyzed (Participants) | 31 | 31
mg of morphine equivalents | 0 [0 to 45] | .5 [0 to 38]

10. Secondary Outcome: Total Opioid Taken by Patient as Tabulated and Converted to Morphine Equivalents
Description: opioid use from time 48-72 hours in mg morphine equivalents
Time Frame: 48-72 hours after end of surgery
Measure: Median (Full Range); unit: mg morphine equivalents
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
Number analyzed (Participants) | 31 | 31
mg morphine equivalents | 0 [0 to 25] | 5 [0 to 34]

11. Secondary Outcome: Patient Satisfaction With Pain Management
Description: number of patients who answered yes to if they were satisfied with their pain management
Time Frame: at 72 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
Number analyzed (Participants) | 31 | 31
Participants | 30 | 24

12. Secondary Outcome: Maximal Pain Score of Patient From Time 0-24 Hours After Surgery
Description: the maximal pain score felt by patient during this time period. This is based on a numerical rating scale of 0-10. 0 is best outcome and 10 is worst outcome.
Time Frame: 0-24 hours after surgery
Measure: Median (Full Range); unit: units on a scale
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
Number analyzed (Participants) | 31 | 31
units on a scale | 3 [0 to 10] | 5 [2 to 10]

13. Secondary Outcome: Maximal Pain Score for Patient From Time 24-48 Hours After Surgery
Description: as for outcome 12
Time Frame: 24-48 hours after surgery
Measure: Median (Full Range); unit: units on a scale
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
Number analyzed (Participants) | 31 | 31
units on a scale | 3 [0 to 9] | 4 [0 to 10]

14. Secondary Outcome: Maximal Pain Score Patient Felt From 48-72 Hours After Surgery
Description: as for outcome 12
Time Frame: 48-72 hours after surgery
Measure: Median (Full Range); unit: units on a scale
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
Number analyzed (Participants) | 31 | 31
units on a scale | 2 [0 to 10] | 3 [0 to 10]

ADVERSE EVENTS:
Time Frame: adverse event data was kept up to 30 days after surgery
Arm/Group | TAP-Block With Liposomal Bupivacaine | Surgical Infiltration With Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 10/31 | 16/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAP-Block With Liposomal Bupivacaine (N=31) | Surgical Infiltration With Bupivacaine (N=31)
nausea/vomiting (Gastrointestinal disorders) | 10 (10) | 16 (16) — number of patients who had nausea/vomiting after surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2015-07-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT02519023/Prot_000.pdf